CLINICAL TRIAL: NCT00107900
Title: A Phase IIa, Multi-center, Multi-national, Open Label, Dose Ranging Study of the Efficacy, Safety, and Tolerability of Oral DU-176b Administered Once or Twice Daily in the Treatment of Adult Patients Undergoing Total Hip Arthroplasty
Brief Title: Study of the Efficacy and Safety of DU-176b in Preventing Blood Clots in Patients Undergoing Total Hip Replacement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Anne MacDonald, Daiichi Sankyo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DU176b-PRT007
Record Dates: First submitted 2005-04-11; First posted 2005-04-12 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2015-02

CONDITIONS: Arthroplasty, Replacement, Hip; Thrombosis
Keywords: Deep Vein Thrombosis,; Anticoagulant,; Venous thromboembolic
MeSH Terms: conditions — Thrombosis; Venous Thrombosis | interventions — edoxaban

ARMS (6):
- 15mg BID (Experimental): 15mg edoxaban administered twice daily (BID)
  Interventions: Drug: DU-176b
- 30mg QD (Experimental): 30mg edoxaban administered once daily (QD)
  Interventions: Drug: DU-176b
- 30mg BID (Experimental): 30mg edoxaban administered twice daily (BID)
  Interventions: Drug: DU-176b
- 60mg QD (Experimental): 60mg edoxaban administered once daily (QD)
  Interventions: Drug: DU-176b
- 60mg BID (Experimental): 60mg edoxaban administered twice daily (BID)
  Interventions: Drug: DU-176b
- 120mg QD (Experimental): 120mg edoxaban administered once daily (QD)
  Interventions: Drug: DU-176b

INTERVENTIONS:
Drug: DU-176b

SUMMARY:
Patients who undergo total hip replacement surgery are at greater risk of getting deep vein thrombosis (blood clots). This study evaluates the safety, tolerability and effectiveness of the study drug, DU-176b, in reducing the occurrence of deep vein thrombosis in patients having total hip replacement surgery.

DETAILED DESCRIPTION:
The primary study objective is to demonstrate prevention of venous thromboembolism in patients undergoing total hip replacement surgery. The secondary objective is to assess the safety and tolerability of DU-176.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral hip replacement

Exclusion Criteria:

* Patients scheduled for bilateral hip replacement in same procedure
* Patients with increased risk of bleeding
* Uncontrolled hypertension (BP greater than 180/100 mmHg)
* Patients less than 111 lbs or more than 243 lbs
* Patients on long-term anticoagulants
* Patients with contraindications to venography
* Patients with medical history of venous thromboembolism
* Patients with impaired hepatic function
* Known to be pregnant
* Lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2005-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Local Institution, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 15mg BID | 30mg QD | 30mg BID | 60mg QD | 60mg BID | 120mg QD
Started | 85 | 75 | 129 | 99 | 115 | 103
Completed | 75 | 72 | 104 | 87 | 94 | 94
Not Completed | 10 | 3 | 25 | 12 | 21 | 9
Not completed — Adverse Event | 3 | 2 | 10 | 3 | 5 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 4 | 1 | 3 | 2 | 5 | 5
Not completed — Protocol Violation | 1 | 0 | 5 | 5 | 7 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 5 | 0 | 1 | 1
Not completed — Administrative Reasons | 1 | 0 | 2 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15mg BID | 30mg QD | 30mg BID | 60mg QD | 60mg BID | 120mg QD | Total
Number analyzed (Participants) | 85 | 75 | 129 | 99 | 115 | 103 | 606
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (10.71) | 59.0 (11.06) | 60.1 (13.09) | 58.6 (11.90) | 58.8 (12.80) | 56.5 (12.83) | 58.5 (12.25)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 48 | 73 | 65 | 78 | 72 | 396
  >=65 years | 25 | 27 | 56 | 34 | 37 | 31 | 210
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 48 | 71 | 62 | 69 | 56 | 350
  Male | 41 | 27 | 58 | 37 | 46 | 47 | 256
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 12 | 0 | 3 | 3 | 19
  White | 84 | 75 | 115 | 97 | 108 | 99 | 578
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 1 | 4 | 0 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 6 | 2 | 4 | 0 | 12
  Not Hispanic or Latino | 20 | 11 | 83 | 22 | 31 | 27 | 194
  Unknown or Not Reported | 65 | 64 | 40 | 75 | 80 | 76 | 400
Region of Enrollment [Number; unit: participants]
  United States | 20 | 11 | 89 | 24 | 35 | 27 | 206
  Europe | 65 | 64 | 40 | 75 | 80 | 76 | 400

OUTCOME MEASURES:

1. Primary Outcome: Prevention of Venous Thromboembolism (VTE)
Description: The primary efficacy endpoint was the proportion of subjects who experienced at least one of the thromboembolic events listed below during the period from the start of study treatment to the venography at the end of study treatment (approximately 2 weeks post surgery).
  Confirmed deep vein thrombosis ( both proximal and distal ) as assessed by unilateral or bilateral ascending contrast venograms 7 to 10 days following surgery Symptomatic and objectively proven Pulmonary Embolism (PE) prior to venography Symptomatic and objectively proven Deep Vein Thrombosis (DVT) prior to venography
Time Frame: 2 weeks
Population: modified ITT population
Measure: Number (90% Confidence Interval); unit: percentage of patients with event
Arm/Group | 15mg BID | 30mg QD | 30mg BID | 60mg QD | 60mg BID | 120mg QD
Number analyzed (Participants) | 68 | 65 | 97 | 73 | 84 | 80
percentage of patients with event | 13 [11.7 to 28.7] | 13 [12.3 to 29.9] | 10 [5.7 to 16.9] | 13 [10.9 to 26.8] | 16 [12.3 to 27.5] | 17 [14.0 to 30.2]
Statistical Analysis 1: Comparison: 15mg BID vs 30mg QD vs 30mg BID vs 60mg QD vs 60mg BID vs 120mg QD; Test type: Superiority or Other; p = 0.238, Fisher Exact

2. Secondary Outcome: Change From Baseline for Prothrombin Time (PT) Results
Description: Intent to Treat (ITT) population
Time Frame: end of treatment
Population: ITT population
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 15mg BID | 30mg QD | 30mg BID | 60mg QD | 60mg BID | 120mg QD
Number analyzed (Participants) | 72 | 72 | 86 | 84 | 95 | 91
seconds | -.2 (2.3) | -.1 (2.7) | .7 (1.3) | .8 (2.0) | 1.1 (1.9) | 1.8 (4.3)

3. Secondary Outcome: Change From Baseline for International Normalized Ratio (INR) Results
Description: Intent to Treat (ITT) population
Time Frame: end of treatment
Population: ITT population
Measure: Mean (Standard Deviation); unit: INR ratio
Arm/Group | 15mg BID | 30mg QD | 30mg BID | 60mg QD | 60mg BID | 120mg QD
Number analyzed (Participants) | 72 | 72 | 86 | 84 | 95 | 91
INR ratio | 0 (.2) | 0 (.3) | .1 (.1) | .1 (.2) | .1 (.2) | .2 (.4)

4. Secondary Outcome: Change From Baseline for Activated Partial Thromboplastin Time (aPTT) Results
Description: Intent to Treat (ITT) population
Time Frame: end of treatment
Population: ITT population
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 15mg BID | 30mg QD | 30mg BID | 60mg QD | 60mg BID | 120mg QD
Number analyzed (Participants) | 72 | 72 | 87 | 84 | 94 | 91
seconds | -5.1 (22.0) | -1.6 (25.3) | 2.5 (9.8) | 4.1 (17.0) | 5.8 (16.1) | 11.3 (23.1)

ADVERSE EVENTS:
Arm/Group | 15mg BID | 30mg QD | 30mg BID | 60mg QD | 60mg BID | 120mg QD
Serious Adverse Events (participants affected / at risk) | 4/85 | 3/75 | 9/129 | 10/99 | 10/115 | 4/103
Other Adverse Events (participants affected / at risk) | 24/85 | 19/75 | 65/129 | 56/99 | 66/115 | 34/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15mg BID (N=85) | 30mg QD (N=75) | 30mg BID (N=129) | 60mg QD (N=99) | 60mg BID (N=115) | 120mg QD (N=103)
obstructive inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
haematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
blood alkaline phosphatase abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
alanine aminotransferase abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
blood bilirubin abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
aspartate amniotransferase abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hepatic enzyme increase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
sciatic nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
snake bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
contrast media reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
wound haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
postprocedural fistula (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
acute psychosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
anemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
lymphadentis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
hip arthroplasty (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
alanine aminotransferase increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
blood alkaline phosphatase increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
anxiety (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 15mg BID (N=85) | 30mg QD (N=75) | 30mg BID (N=129) | 60mg QD (N=99) | 60mg BID (N=115) | 120mg QD (N=103)
tachycardia (Cardiac disorders) | 1 | 1 | 1 | 7 | 3 | 3
constipation (Gastrointestinal disorders) | 3 | 4 | 24 | 7 | 12 | 8
nausea (Gastrointestinal disorders) | 3 | 2 | 9 | 6 | 8 | 4
hyperthermia (General disorders) | 8 | 5 | 5 | 27 | 23 | 9
oedema peripheral (General disorders) | 6 | 3 | 12 | 4 | 11 | 5
pyrexia (General disorders) | 3 | 4 | 23 | 10 | 11 | 9
procedural pain (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 3 | 6 | 0
activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 13 | 5 | 6
prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 15 | 3 | 4
dizziness (Nervous system disorders) | 1 | 0 | 7 | 4 | 3 | 1
headache (Nervous system disorders) | 0 | 1 | 9 | 1 | 4 | 2
insomnia (Psychiatric disorders) | 0 | 0 | 9 | 5 | 5 | 0
anaemia (Blood and lymphatic system disorders) | 2 | 3 | 8 | 2 | 10 | 8
anaemia post-operative (Injury, poisoning and procedural complications) | 3 | 1 | 5 | 5 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A study site may not publish results of a study until after a coordinated multicenter publication has been submitted for publication or until one year after the study has ended, whichever occurs first. The study site will have the opportunity to publish results of the study, provided Daiichi Sankyo has had the opportunity to review and comment on the study site's proposed publication prior to being submitted for publication with the advice of patent council and need for subject protection.